CLINICAL TRIAL: NCT06521684
Title: Translational Study of MSS, TP53 Mutation and Chromosome Instability Relationship in Endometrial Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECMTC
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Neoplasms; TP53 Gene Mutation; Chromosomal Instability; Microsatellite Stable Endometrial Carcinoma
Keywords: Endometrial Cancer; Chromosomal Instability; microsatellite stability; TP53 Gene Mutation; Whole genome duplication
MeSH Terms: conditions — Endometrial Neoplasms; Chromosomal Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Preserved or fresh tumor tissue. Tumor tissue samples were embedded in paraffin wax, section thickness was 6μm, and section number was 10 (surgical tissue) or 15 (puncture tissue). Tumor cell content > 30%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to understand the relationship between TP53 mutation, MSS and chromosome instability in endometrial cancer and the effect on clinical prognosis.We will collect a small amount of tumor tissue samples. NGS panel detection and WGD/AS analysis were performed on the tissue. Paracancer tissue was used as a negative control and relevant information in medical records during the operation. Then we will collect clinical diagnosis and disease information through telephone follow-up after the completion of the operation.

DETAILED DESCRIPTION:
The test is sequenced using Illumina high-throughput sequencers and accompanying kits. Conduct preliminary quality control on the samples, and the tumor cell content of the tissue samples shall not be less than 30%. Tissue DNA was extracted from tumor tissue samples according to the instructions of the QIAGEN DNA extraction kit. Samples qualified for quality control shall be arranged for further library construction. The extracted DNA samples were sequentially purified by fragment purification, terminal repair, splicing, fragment size selection, PCR amplification, product purification, library enrichment, and library product quality control. After qualified quality control, the constructed library was sequenced by Illumina matching kit. Bioinformatics analysis would be conducted.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study and sign the informed consent
* age ≥18 years old
* researchers evaluated that it was suitable to participate in this translational study
* Endometrial cancer was confirmed histologically
* histopathological molecular classification was consistent with pMMR type and POLE wild type
* The tumor tissue obtained by operation was the primary lesion

Exclusion Criteria:

* Received chemotherapy within 14 days prior to sample collection, or received anti-tumor drug therapy such as radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, within 21 days prior to sample collection
* previously treated with KIF18A inhibitors
* researchers believed that the subjects were not suitable for the translational study for other reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective and retrospective samples were collected from September 1, 2024 to June 30, 2025, with an estimated total sample size of 110 cases, including 80 fresh tumor tissues and 30 archival tumor tissues. There were 40 TP53 mutations (high copy type) and 70 TP53 negative (MSS type).
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
microsatellite stability status | 2025-06-30
  microsatellite stability status
TP53 mutation | 2025-06-30
  TP53 mutation
Chromosomal instability | 2025-06-30
  Chromosomal instability (Whole genome duplication, Aneuploidy)

SECONDARY OUTCOMES:
recurrence | 2026-06-30
  disease recur